CLINICAL TRIAL: NCT05057845
Title: A Phase II Study of Cryoablation Combined with Tislelizumab Plus Lenvatinib As Second-line or Later Therapy in Patients with Advanced Hepatocellular Carcinoma (CASTLE-02)
Brief Title: Cryoablation Combined with Tislelizumab Plus Lenvatinib As Second-line or Later Therapy in Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Peng Wang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASTLE-02
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — tislelizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cryoablation in combination with Tislelizumab plus lenvatinib (Experimental)
  Interventions: Drug: Tislelizumab; Drug: lenvatinib; Combination Product: US/CT-guided Percutaneous Cryoablation

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab will be initiated on day 14 after cryoablation. Tislelizumab will be administered at 200 mg i.v. every 3 weeks
Drug: lenvatinib — Lenvatinib will be initiated on day 14 after cryoablation. Lenvatinib will be administered (bodyweight ≥ 60 kg, 12 mg; < 60 kg, 8 mg) orally daily every 3 weeks until documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
Combination Product: US/CT-guided Percutaneous Cryoablation — Cryoablation will be performed with a two-cycle freeze-thaw phase protocol; US or non-contrast CT images will be obtained to visualize the evolving ablation zone

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of cryoablation combined with Tislelizumab plus lenvatinib as second-line or later therapy in patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
Recent studies have suggested that local destruction of tumor tissue by cryoablation induced activation and maturation of dendritic cells and tumor-specific T cells by cross-presentation of tumor antigens. While pd-1 blocking antibody interferes with PD-1 mediated T-cell regulatory signaling. And combination of pd-1 blocking antibody plus lenvatinib showed increased ORR in many type of human cancers, including advanced hepatocellular carcinoma. Therefore, the objective of this study is to evaluate the efficacy and safety of cryoablation combined with Tislelizumab plus lenvatinib as second-line or later therapy in patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Age ≥ 18 years at time of study entry.
* Participants must have unresectable or metastatic histologically or cytologically confirmed hepatocellular carcinoma
* Participants must have failed 1 line of systemic regimens for advanced hepatocellular carcinoma due to disease progression or toxicity.
* Patients had been refractory or intolerant to previous systemic chemotherapy (oxaliplatin-based chemotherapy), targeted therapy (eg, sorafenib or lenvatinib), or anti-PD-1 or anti-PD-L1 based regimen.
* At least one measurable site of disease as defined by RECIST criteria with spiral CT scan or MRI.
* Performance status (PS) ≤ 2 (ECOG scale).
* Life expectancy of at least 12 weeks.
* Adequate blood count, liver-enzymes, and renal function: absolute neutrophil count ≥ 1,500/L, platelets ≥75 x103/L; Total bilirubin ≤ 3x upper normal limit; Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT) ≤ 5 x upper normal limit (ULN); International normalized ratio (INR) ≤1.25; Albumin ≥ 31 g/dL; Serum Creatinine ≤ 1.5 x institutional ULN or creatinine clearance (CrCl) ≥ 30 mL/min (if using the Cockcroft-Gault formula )
* Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment, adherence to contraceptive measures, scheduled visits and examinations including follow up.

Exclusion Criteria:

* History of cardiac disease, including clinically significant gastrointestinal bleeding within 4 weeks prior to start of study treatment
* Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months Prior to the first dose of study drug with the exception of thrombosis of a segmental portal vein.
* Prior treatment with cryoablation.
* RFA and resection administered less then 4 weeks prior to study treatment start.
* Radiotherapy administered less then 4 weeks prior to study treatment start.
* Major surgery within 4 weeks of starting the study treatment OR subjects who have not recovered from effects of major surgery.
* Patients with second primary cancer, except adequately treated basal skin cancer or carcinoma in-situ of the cervix.
* Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is longer.
* Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study Treatment or interpretation of patient safety or study results, including but not limited to:

  1. history of interstitial lung disease
  2. Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) coinfection (i.e double infection)
  3. known acute or chronic pancreatitis
  4. active tuberculosis
  5. any other active infection (viral, fungal or bacterial) requiring systemic therapy
  6. history of allogeneic tissue/solid organ transplant
  7. diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of Tislelizumab treatment.
  8. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions: Subjects with vitiligo, hypothyroidism, diabetes mellitus type I or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with Hashimoto thyroiditis, hypothyroidism stable on hormone replacement or psoriasis not requiring treatment are not excluded from the study.
  9. Live vaccine within 30 days prior to the first dose of Tislelizumab treatment or during study treatment.
  10. History or clinical evidence of Central Nervous System (CNS) metastases Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria: I. are asymptomatic and II. have no requirement for steroids 6 weeks prior to start of Tislelizumab treatment. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS
* Medication that is known to interfere with any of the agents applied in the trial.
* Any other efficacious cancer treatment except protocol specified treatment at study start.
* Patient has received any other investigational product within 28 days of study entry.
* Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (serum β-HCG) at screening.
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-09-26 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | max 24 months
  ORR according to RECIST 1.1

SECONDARY OUTCOMES:
DoR | max 24 months
  Duration of Response
PFS | max 24 months
  Progression Free Survival
OS | max 42 months
  Overall survival
DCR | max 24 months
  disease control rate
Adverse Events | max 42 months
  Adverse event (AE)、Treatment emergent adverse event(TEAE)、Serious adverse event (SAE).

CONTACTS AND LOCATIONS:
Overall Officials: Peng Wang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China